CLINICAL TRIAL: NCT01086813
Title: Phase I, Single Centre, Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous AZD3043 After a Single Ascending Bolus Dose Followed by a Single Infusion Dose in Elderly (=65 Years) Healthy Volunteers
Brief Title: Phase I, Single Centre, Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD3043
Acronym: AZD3043
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The compound is being re-evaluated
Sponsor: AstraZeneca (Industry)
Responsible Party: AstraZeneca, AstraZeneca
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D0510C00005; AZD3043
Record Dates: First submitted 2010-03-09; First posted 2010-03-15 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Safety; Tolerability; Pharmacokinetics; Sedation
Keywords: Safety; Tolerability; Pharmacokinetics; Sedation
MeSH Terms: interventions — AZD-3043

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD3043

INTERVENTIONS:
Drug: AZD3043 — single dose/IV, bolus over 60secs - infusion over 30 mins

SUMMARY:
Phase I, Single Centre, Open Label Study to Assess the Safety, Tolerability,Pharmacokinetics and Pharmacodynamics of Intravenous AZD3043 after aSingle Ascending Bolus Dose Followed by a Single Infusion Dose in Elderly(=65 years) Healthy Volunteers

DETAILED DESCRIPTION:
Phase I, Single Centre, Open Label Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenous AZD3043 after a Single Ascending Bolus Dose Followed by a Single Infusion Dose in Elderly (=65 years) Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Pre-anaesthesia assessment judged without remarks by the investigator.
* ASA physical status category 1 to 2 (up to and including 3 depending on applicable patient category)

Exclusion Criteria:

* Lack of a normal range of enzyme activity for BuChE
* Known or suspected history of hypersensitivity to drugs with a similar chemical structure or class to AZD3043 (e.g., emulsion-based products like Diprivan,Intralipid), allergies to soybean or peanut products or any other drugs intended for use during th
* Prolonged QTcF >450 ms or shortened QTcF <350 ms or family history of long QT syndrome.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-03; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability after administration of a bolus and infusion of AZD3043 | Heartrate, Bloodpressure, Telemetry, ECG, EtCO2, SPO2, BIS, Respiratory frequency every minute during a 1h session

SECONDARY OUTCOMES:
To evaluate the PK of AZD3043 and its main metabolite (THRX-108893) in venous blood samples | During 24h
To evaluate the onset, level and recovery from sedation/anaesthesia | During 24h

CONTACTS AND LOCATIONS:
Overall Officials: Darren Wilbraham, Principal Investigator — Quintiles Drug Research Unit at Guy's HospitalQuintiles Ltd6 Newcomen StreetLondonSE1 1YRUnited Kingdom; Stephen Kanes, Study Director — AstraZeneca; Brendan Smyth, Study Chair — AstraZeneca